CLINICAL TRIAL: NCT00003197
Title: Phase I Evaluation of Green Tea Extract in Adults With Advanced Solid Tumors
Brief Title: Green Tea Extract in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-128; CDR0000066033 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1375
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Tea

INTERVENTIONS:
Dietary Supplement: green tea extract

SUMMARY:
RATIONALE: Green tea extract contains ingredients that may slow the growth of certain cancers, as well as prevent the development of new cancers.

PURPOSE: Phase I trial to study the effectiveness of green tea extract in treating patients with advanced solid tumors that are refractory to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of green tea extract administered daily to adults with solid tumors. II. Determine the safety of chronic daily administration of green tea extract in these patients. III. Investigate the clinical pharmacology of green tea extract in this study. IV. Document observed antitumor activity of this treatment.

OUTLINE: This is a dose escalation study of green tea extract. Patients receive green tea extract by mouth daily after meals for 4 weeks. One patient is entered at each dose level. If grade II toxicities are experienced, then 2 more patients are entered at the same dose level. One patient must complete 4 weeks of therapy and 2 others must complete 2 weeks of therapy with no greater than grade I toxicity before dose escalation proceeds. If at least 2 patients experience dose limiting toxicity at any dose level, the immediately preceding dose level is considered the maximum tolerated dose (MTD). At least 6 patients are studied at the MTD. Patients may continue therapy for up to 6 months in the absence of toxicity and disease progression. Patients are followed every 4 weeks for the duration of treatment and at least one month after completing treatment.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically proven incurable advanced solid tumor refractory to standard therapy or for which no standard therapy exists No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 OR Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST less than 1.25 times normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No significant cardiac disease Other: No significant metabolic disorder No significant infection Not pregnant or nursing Effective contraception must be used by fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks (6 weeks for nitrosourea) since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-12; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent A. Miller, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States